CLINICAL TRIAL: NCT03925558
Title: Tolerance of a Probiotic Formula Containing Lactobacilli
Brief Title: Tolerance of a Probiotic Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ProTolerance
Record Dates: First submitted 2019-04-17; First posted 2019-04-24 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Safety Issues
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic formula (Active Comparator): Lactobacillus strains
  Interventions: Dietary Supplement: Probiotics
- Placebo formula (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics
  Arms: Probiotic formula
Dietary Supplement: Placebo
  Arms: Placebo formula

SUMMARY:
Evaluate the tolerance of a probiotic formula in infants

ELIGIBILITY:
Inclusion Criteria:

- Full term healthy infant aged 3-95 days

Exclusion Criteria:

* Prematurity
* Low birth weight
* Congenital anomalies
* Chronic disease
* Failure to thrive
* Allergy or atopic disease
* Recent exposure to antibiotics

Ages: 3 Days to 95 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2011-04-12 (Actual); Primary Completion 2011-12-19 (Actual); Study Completion 2011-12-19 (Actual)

PRIMARY OUTCOMES:
Body weight (g) | 8 weeks
Body length (cm) | 8 weeks
Head circumference (cm) | 8 weeks

IPD SHARING:
Plan to Share IPD: No